CLINICAL TRIAL: NCT02634099
Title: Hemoglobin Monitoring During High Bleeding Risk Surgery in Pediatric Patients: Equivalence Study of Hemoglobin Transcutaneous Saturation and Hemocue With Total Serum Hemoglobin
Brief Title: A Comparison of Three Methods of Hemoglobin Monitoring in Pediatric Patients Undergoing Major Surgery
Acronym: Hemoped
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-A00916-43
Record Dates: First submitted 2015-12-08; First posted 2015-12-17 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Child
Keywords: major pediatric surgery; hemoglobin measurement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- hemoglobine monitoring (Other): 3 different techniques will be used for hemoglobine monitoring : hemocue, pulse co-oxymeter (SpHb) and blood measurement
  Interventions: Device: blood measurement; Device: pulse co-oxymeter (SpHb); Device: hemoCue

INTERVENTIONS:
Device: blood measurement — Hemoglobin measurement
Device: pulse co-oxymeter (SpHb) — non invasive method of hemoglobin measurement
Device: hemoCue — non invasive method of hemoglobin measurement

SUMMARY:
Investigators compare the accuracy of the SpHb and hemocue with blood Hb levels

DETAILED DESCRIPTION:
The goal of the study is to compare 3 methods of hemoglobin measurement in pediatric patients undergoing major surgery. During general anesthesia investigators will measure and compare at different periods of time blood hemoglobin levels obtained from a radial artery catheter with 2 non invasive methods of measurement using hemocue and SpHb

ELIGIBILITY:
Inclusion Criteria:

Paediatric patients scheduled for major orthopaedi or neurosurgical process under general anesthesia Arterial catheter necessary in the anesthetic protocol. BMI<30 No opposition holders of parental authority and children.

Exclusion Criteria:

Hemoglobin disease Pretreatment with erytropoietin or iron

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2016-01-05 (Actual); Primary Completion 2016-11-23 (Actual); Study Completion 2016-11-23 (Actual)

PRIMARY OUTCOMES:
comparison of hemoglobin measurement using 3 different techniques at the time of transfusion decision | within the day of surgery
  comparison of blood hemoglobin obtained by arterial samples with 2 non invasive methods of measurement using hemocue and SpHb

CONTACTS AND LOCATIONS:
Overall Officials: Claude MEISTELMAN, MD, Principal Investigator — CHRU NANCY
Locations (1):
- Chru Nancy, Vandœuvre-lès-Nancy, France